CLINICAL TRIAL: NCT00291902
Title: A 28-day, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Anti-inflammatory Effect and Steady-state Pharmacokinetics of SB-681323 (7.5 mg) in Subjects With Coronary Heart Disease (CHD) Undergoing Elective Percutaneous Coronary Interventions (PCI)
Brief Title: A Pharmacokinetic Study Of SB-681323 In Subjects With Coronary Heart Disease Undergoing Percutaneous Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMK103351
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Heart Disease
Keywords: CHD; coronary heart disease; atherosclerosis; inflammation
MeSH Terms: conditions — Coronary Disease; Atherosclerosis; Inflammation | interventions — dilmapimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-681323

SUMMARY:
Study of SB-681323 (a novel p38 MAPkinase inhibitor) in subjects with documented coronary heart disease (CHD) undergoing elective percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Females must be of non-child-bearing potential.
* Female subjects must have a negative pregnancy test.
* Subjects scheduled to undergo elective single vessel PCI to be performed within the 6 weeks of diagnostic coronary angiography.
* Must be on stable dose of statin for = 6 weeks prior to screening, with statin tolerability and LDL <130 mg/dL (3.4 mmol/L) at Screening visit.
* Must be capable of providing informed consent.
* Have an hsCRP concentration of >2 mg/L, but < 10 mg/L at screening.

Exclusion Criteria:

* Women who are pregnant or breast feeding.
* Planned PCI with multi-vessel stenting.
* Planned PCI with additional revascularization procedures staged at different days during the study period.
* Planned PCI other than stenting (e.g., atherectomy, PTCA without stenting, etc).
* Planned PCI of any bypass graft.
* History of CABG surgery.
* Planned cardiac or major non-cardiac surgery within the study period.
* Disabling stroke in the past 6 months.
* History of chronic viral hepatitis or other chronic hepatic disorders.
* History of Gilbert's syndrome or elevated bilirubin concentrations at screening.
* History of increased liver function tests (ALT, AST) due to acute or chronic liver conditions, above the upper limit of normal at screening or in the past 6 months.
* Renal impairment with serum creatinine >2.0 mg/dl (177umol/L) at Screening, or history of kidney transplant, or a history of contrast nephropathy.
* Current inadequately controlled hypertension (blood pressure >160 mmHg systolic and/or >100 mmHg diastolic) on a stable dose of antihypertensive medication.
* Current poorly controlled diabetes mellitus, defined as HbA1c >10% at Screening.
* History of severe heart failure defined as NYHA class III or IV or those with known severe LV dysfunction (EF<30%) regardless of symptomatic status.
* History of malignancy within the past 5 years, other than non-melanoma skin cancer.
* Current life-threatening condition other than vascular disease that may prevent a subject from completing the study.
* Alcohol or drug abuse within the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-03

PRIMARY OUTCOMES:
Patient safety Tolerability Anti-inflammatory effect (high sensitivity C-reactive Protein) | 28 days

SECONDARY OUTCOMES:
Anti-inflammatory effect (biomarkers) Endothelial function (peripheral artery tonometry) Pharmacokinetics | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Denmark (5):
  - GSK Investigational Site, Esbjerg
  - GSK Investigational Site, Haderslev
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Herning
  - GSK Investigational Site, Viborg
- Poland (2):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Poznan

REFERENCES:
- [Derived] Sarov-Blat L, Morgan JM, Fernandez P, James R, Fang Z, Hurle MR, Baidoo C, Willette RN, Lepore JJ, Jensen SE, Sprecher DL. Inhibition of p38 mitogen-activated protein kinase reduces inflammation after coronary vascular injury in humans. Arterioscler Thromb Vasc Biol. 2010 Nov;30(11):2256-63. doi: 10.1161/ATVBAHA.110.209205. Epub 2010 Aug 5. PMID 20689074